CLINICAL TRIAL: NCT07073625
Title: The Effects of Stress Ball and Storybook Reading During Inhaler Application on Fear and Anxiety in Children
Brief Title: During Inhaler Application, Children Were Given Stress Ball and Storybook Reading Interventions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Zülbiye demir barbak, Lecturer, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Stress Ball, Reading Storybook
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Inhalation Therapy
Keywords: Inhalation therapy; Fear; Anxiety; Stress Ball; Reading Storybook; Child
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine clinical care will be applied to the control group. No action will be taken.
- Experimental Group (Experimental): Children aged 5-6 who come to the emergency room with their parents and will receive inhalers will be given stress ball balls in the stress ball group before and after the procedure and will be told to play with them until the procedure is completed. In the book reading group, parents will be asked to read a book about hospital fear, prepared by researchers.
  Interventions: Other: Stress Ball; Other: Reading Storybook

INTERVENTIONS:
Other: Stress Ball — Children arriving at the hospital's emergency department and meeting the study criteria will be randomly assigned to the stress ball group. Before inhalation therapy, the child will begin squeezing the chosen stress ball. This will distract their attention, transforming the frightening hospital environment into a fun one. The questionnaires will be completed by the nurse and family five minutes before, during, and after the inhalation therapy.
  Arms: Experimental Group
Other: Reading Storybook — The storybook for the children will be selected by child psychologists. The book will be read to the children by their parents. The storybook reading will begin 15 minutes before the inhalation therapy and will be completed before the treatment begins. The storybook will be read to the children only once.
  Arms: Experimental Group

SUMMARY:
It aims to examine the effects of stress ball and book reading methods on children's fear and anxiety levels during inhalation.

DETAILED DESCRIPTION:
Ninety-nine volunteer children aged 5-6 who will receive inhalation therapy will be randomly assigned to three groups: stress ball, storybook reading, and control. Children will be assessed before, during, and after the procedure. Inhalation-related fear will be assessed using the Children's Fear Scale, and anxiety will be assessed using the Children's State Anxiety Scale. Furthermore, children's demographic data will be recorded on the Information Form.

ELIGIBILITY:
Inclusion Criteria:

* No audiovisual impairment,
* Being open to communication and
* Must be accompanied by a parent.

Exclusion Criteria:

* Having special needs,
* Having an audio-visual impairment,
* Learning difficulties or mental retardation and
* Children whose parents do not agree to participate in the study.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Demographic Information Form | Baseline
  It is a form consisting of a total of 13 questions including the child's age, gender, diagnosis, duration of treatment, number of treatments (How many times did the child come to the clinic?), the status of receiving information about dental treatment and the person who received the information, the education level and occupation of the mother and father, the place where the family lives and the economic situation. It was prepared by the researchers in line with the literature.
Child anxiety Scale-State | Baseline and up to 4 weeks
  "Child Anxiety Scale-State" scale developed by Ersig et al. in 2013 measures the state anxiety of children aged 4-10 years. In 2017, Gerceker et al. carried out Turkish validity study for the scale. CAS-S (State) is designed as a thermometer. At the bottom is the bulb chamber, and upward are horizontal lines. Each horizontal line represents a score, and the thermometer has 10 points. The bulb chamber at the bottom is 0 points and indicates that there is no anxiety. It is interpreted as the rise of anxiety as it rises upwards. The peak is worth 10 points and refers to the highest anxiety.
Child Fear Scale | Baseline and up to 4 weeks
  This scale was developed by McMurtry et al. in 2011. In 2018, Gerceker et al. carried out a Turkish validity study for the scale. The scale is aimed at children aged 5-10 years. The facial muscle changes in fearful expressions are drawn by a graphic artist based on photos of frightened faces. In this scale, the child is shown a scale containing five facial expressions that are evaluated between 0 and 4 points. While 0 point refers to no fear; 4 points refers to the highest fear.

CONTACTS AND LOCATIONS:
Overall Officials: Zülbiye DEMİR BARBAK, 1, Principal Investigator — Ataturk University
Locations (1):
- Erzurum City Hospital, Erzurum, Center, Turkey (Türkiye)

REFERENCES:
- [Background] Aminabadi NA, Vafaei A, Erfanparast L, Oskouei SG, Jamali Z. Impact of pictorial story on pain perception, situational anxiety and behavior in children: a cognitive-behavioral schema. J Clin Pediatr Dent. 2011 Winter;36(2):127-32. doi: 10.17796/jcpd.36.2.3163251527508338. PMID 22524072
- See also: Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/22524072/